CLINICAL TRIAL: NCT02839577
Title: The Effect of High Volume Injection With and Without Steroid in Chronic Achilles Tendinopathy: A Randomized Double Blinded Prospective Trial
Brief Title: The Effect of High Volume Injection With and Without Steroid in Chronic Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Anders Ploug Boesen, MD, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: H-1-2010-052b
Record Dates: First submitted 2016-07-08; First posted 2016-07-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Tendinopathy
MeSH Terms: conditions — Tendinopathy | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Volume injection (HVI) with corticosteroid (Active Comparator): * 10 mls 0.5% bupivacaine hydrochloride
  * 20 mg of Depomedrol (40 mg/ml methylprednisolonacetat)
  * 40 mls saline (NaCl)
  HVI with corticosteroid is injected one time at baseline and compared to HVI without corticosteroid.
  Interventions: Drug: High Volume injection without corticosteroid
- High Volume injection (HVI) without corticosteroid (Active Comparator): * 10 mls 0.5% bupivacaine hydrochloride
  * 40 mls saline (NaCl)
  HVI with corticosteroid is injected one time at baseline and compared to HVI with corticosteroid.
  Interventions: Drug: High Volume injection with corticosteroid

INTERVENTIONS:
Drug: High Volume injection without corticosteroid — Injection with 10 mls 0.5% bupivacaine hydrochloride and
  • 40 ml saline around the tendon.
  Other Names: HVI without corticosteroid
  Arms: High Volume injection (HVI) with corticosteroid
Drug: High Volume injection with corticosteroid — Injection with 10 mls 0.5% bupivacaine hydrochloride, 20 mg Depomedrol and 40 ml saline around the tendon.
  Other Names: HVI with corticosteroid
  Arms: High Volume injection (HVI) without corticosteroid

SUMMARY:
The aim of the study is to determine the effect of steroid in High Volume Injection (HVI) compared to HVI without steroid (volume effect) in functional outcomes and ultrasound tendon thickness and Color Doppler activity in chronic Achilles tendinopathy (AT).

Healthy males with AT will be randomly assigned to either 1) HVI with steroid (50 mls;10 mls 0.5% bupivacaine hydrochloride and 20 mg of Depomedrol followed by 40 ml saline) or 2) HVI without steroid (50 mls;10 mls 0.5% bupivacaine hydrochloride followed by 40 ml saline).

All subjects will perform a 12-wk eccentric training program with further eccentric training 3 times per week from week 12 to week 24.

Clinical examinations and ultrasound will be performed at baseline (before treatment) with follow-ups after 6 weeks, 12 weeks and again after 24 weeks prior to baseline to see any possible changes and differences between the two groups.

DETAILED DESCRIPTION:
Chronic Achilles tendinopathy (AT) is a common and impairing disorder. High Volume Injection therapy (HVI) seems to show promising results in Achilles tendinopathy (AT). HVI consist of a large volume of saline with a small amount of steroid. Steroid injections is widely used for treating tendinopathy but we know from the literature that steroid injections only gives a fast and short term pain reduction in tendinopathy where HVI seems to show both a short term and a more prolonged effect which could contribute the volume effect (saline).

Aim: The aim of the study is to determine the effect of steroid in High Volume Injection (HVI) compared to HVI without steroid (volume effect) in functional outcomes and ultrasound tendon thickness and Color Doppler activity in chronic Achilles tendinopathy (AT).

Materials and methods: Healthy males (21-59 years; n=60) with AT is randomly assigned to either 1) HVI with steroid (50 mls;10 mls 0.5% bupivacaine hydrochloride and 20 mg of Depomedrol followed by 40 mls saline) or 2) HVI without steroid (50 mls;10 mls 0.5% bupivacaine hydrochloride followed by 40 mls saline) The injections will be performed under ultrasound guidance. All subjects will undergo a 12 week eccentric training program and the subjects will continue eccentric training 3 times per week from week 12 to week 24.

Clinical effects will be assessed as changes in symptoms and pain (VISA-A and VAS score), tendon ultrasound thickness and color Doppler. All outcome measures will be recorded at baseline and again at 6 weeks, 12 weeks and 24 weeks follow-up.

Statistics: All data will be analyzed in SigmaPlot v11 using two-way repeated measures ANOVA with Student-Newman-Keuls Post-hoc test. This is used to see changes over time in all groups (time effect) and differences between groups within time-points (group effect). All data will be presented as mean ± SEM time.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and ultrasound diagnosed unilateral mid-tendinous Achilles tendinopathy.
* Symptoms > 3 month

Exclusion Criteria:

* Bilateral achilles tendinopathy
* Insertional tendinopathy
* Steroid injections < 12 month
* Diabetes or cardiovascular disease
* Smoking
* Treatment with fluoroquinolones < 6 month

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The Victorian Institute of Sports Assessment-Achilles questionnaire (VISA-A score) | Baseline, 6 weeks, 12 weeks and 24 weeks
  Changes in VISA-A score over time between the two groups

SECONDARY OUTCOMES:
The Visual analogue pain scale (VAS score) | Baseline, 6 weeks, 12 weeks and 24 weeks
  Changes in VAS score over time between the two groups
Ultrasound tendon thickness and color Doppler | Baseline, 6 weeks, 12 weeks and 24 weeks
  Changes in tendon thickness and color Doppler between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sportsmedicine, Bispebjerg hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No